CLINICAL TRIAL: NCT01634672
Title: Prevalence of Gastroesophageal Reflux Disease in Peritoneal Dialysis and Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Song Kyung Ho (Other)
Responsible Party: Sponsor-Investigator, Song Kyung Ho, assistant professor, Konyang University Hospital
Organization: Konyang University Hospital (Other)
Other Study IDs: GERD
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; peritoneal dialysis; hemodialysis
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- hemodialysis patients
- Peritoneal dialysis patients

SUMMARY:
The purpose of this study is to determine the prevalence of GERD among chronic kidney disease with peritoneal dialysis and hemodialysis in Korea.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a common upper gastrointestinal disorder in chronic kidney disease. But, little is known about the prevalence in dialysis patients. The aims of this study were to determine the prevalence of GERD among chronic kidney disease with peritoneal dialysis and hemodialysis in Korea.

ELIGIBILITY:
Inclusion Criteria:

* peritoneal dialysis and hemodialysis patients

Exclusion Criteria:

* a history of abdominal surgery or with a proton pump inhibitor before 1 month and a eradication of H. pylori were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic kidney disease undergoing peritoneal dialysis and hemodialysis over 1 year were enrolled
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of GERD among chronic kidney disease with peritoneal dialysis and hemodialysis | 2 yrs

SECONDARY OUTCOMES:
risk factor for GERD in peritoneal dialysis and hemodialysis patients | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Hyun jung Song, Bechelor's, Principal Investigator — Konyang University Hospital
Locations (1):
- Konyang Univ.Hospital, Daejeon, South Korea